CLINICAL TRIAL: NCT03611491
Title: A Prospective, Open Label, Multicenter, Post Market Study Evaluating Princess® FILLER Lidocaine for the Correction of Nasolabial Folds
Brief Title: Post Market Study Evaluating Princess Filler Lidocaine for the Correction of Nasolabial Folds
Acronym: FINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPH-401-201324
Record Dates: First submitted 2017-11-30; First posted 2018-08-02 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2018-01

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Princess® FILLER Lidocaine (Experimental): Princess FILLER Lidocaine injections up to 10 ml given to the patients at baseline time point
  Interventions: Device: Princess FILLER Lidocaine

INTERVENTIONS:
Device: Princess FILLER Lidocaine — Princess FILLER Lidocaine injection up to 10 ml given to the patients at baseline time point. After 2 week a touch up is given in case to be consider necessary.

SUMMARY:
In this study, eligible subjects with moderate to severe nasolabial folds will be treated with Princess® FILLER Lidocaine and will return for follow-up assessments 2, 4, 24 and 36 weeks after the treatment. A Touch-up treatment may be done at Week 2, if deemed appropriate by the investigator

DETAILED DESCRIPTION:
A prospective, open label, multicenter, post-market investigation. Following informed consent and screening, eligible subjects with moderate to severe nasolabial folds were treated with Princess® FILLER Lidocaine, and were to return for follow-up assessments 2, 4, 24 and 36 weeks after the initial treatment. A Touch-up treatment may be done at Week 2 after initial treatment, if deemed appropriate by the investigator. The performance of the investigational device evaluated by the investigator by assessing severity of nasolabial folds using the Nasolabial Folds Severity Rating Scale (NLF-SRS) (4, 24 and 36 weeks after the initial treatment and in comparison to Day 0) and global aesthetic improvement (4, 24 and 36 weeks after the initial treatment). The subject evaluated pain intensity associated with the treatment (at Day 0 and at Week 2 after initial treatment (if Touch-up treatment occurred)), and satisfaction with the treatment 4, 24 and 36 weeks after the initial treatment.

The safety was evaluated based on occurrence of adverse events, which were collected throughout the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Presence of two fully visible, approximately symmetrical nasolabial folds, with each of the folds scored 2-3 according to the 5-grade NLF-SRS as assessed by the investigator
3. Healthy skin in the facial area and free of diseases that could interfere in cutaneous aging evaluation
4. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation
5. Written signed and dated informed consent

Exclusion Criteria:

Subjects meeting any of the following criteria should not be enrolled:

1. Pregnancy, lactation, planned pregnancy or unwillingness to use contraception at any time during the study (for women of child-bearing potential only)
2. History of mental disorders or emotional instability
3. History of allergic reaction or hypersensitivity to hyaluronic acid, lidocaine, or any amide-based anaesthetic
4. Presence of silicone implant or another non-absorbable substance (permanent fillers) in the nasolabial region
5. Facial surgery or implantation of dermal fillers, absorbable and non-absorbable sutures, laser therapy, dermabrasion, or botulinum toxin application in the nasolabial region within previous twelve months, or chemical peeling within previous three months, or planning to undergo such procedures in the treatment area during the study
6. Presence of infectious, inflammatory, or proliferative lesions in the nasolabial region
7. Cutaneous lesions in the treatment area
8. Known human immune deficiency virus-positive individuals
9. History of allergies against aesthetic filling products and recurrent herpes simplex
10. Tendency to hypertrophic scars, keloid formation and/or pigmentation disorders
11. History or presence of any autoimmune or connective tissue disease, or current treatment with immune therapy
12. Diabetes mellitus or uncontrolled systemic diseases
13. Use of anticoagulant, antiplatelet or thrombolytic medication from ten days pre- to three days post injection
14. Any medical condition which, in the investigator's opinion, prohibits the inclusion in the study
15. Current or previous (within 30 days of enrolment) treatment with another investigational drug and/or medical device or participation in another clinical study
16. Previous enrolment in this clinical investigation
17. Subjects whose participation in clinical trials is prohibited by the Austrian Medical Devices Act (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - MÄZ WIEN Medizinisch Ästhetisches Zentrum Wien, Vienna
  - Yuvell, Vienna

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Nasolabial Folds
Period: Overall Study
Arm/Group | Princess® FILLER Lidocaine
Started | 60; 120 Nasolabial Folds
Completed | 59; 118 Nasolabial Folds
Not Completed | 1; 2 Nasolabial Folds
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Nasolabial Fold
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Number analyzed (Nasolabial Fold) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 60
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 60
Average Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade by Investigator [Mean (Standard Deviation); unit: score on a scale] — The left and right nasolabial folds were graded separately by the investigator on the 5-point Nasolabial Folds-Severity Rating Scale (NLF-SRS) then the average of the two sides was used for analysis. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
  score on a scale | 2.72 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade Based on Investigator Assessment at Week 24
Description: Change from baseline in average Nasolabial Folds-Severity Rating Scale (NLF-SRS) grade based on investigator assessment at week 24 after the initial treatment. The left and right nasolabial folds were graded separately on the 5-point NLF-SRS then the average of the two sides was used for analysis. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
Time Frame: Baseline and Week 24
Population: The population used consists of all participants who received the investigational device and had at least one post-treatment assessment (e.g., first pain assessment after injection). Only subjects with available data for week 24 were included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Nasolabial Fold
Groups:
- Princess® FILLER Lidocaine: Princess FILLER Lidocaine injections up to 10 ml given to the patients at baseline time point
  Princess FILLER Lidocaine: Princess FILLER Lidocaine injection up to 10 ml given to the patients at baseline time point. After 2 week a touch up is given in case to be considered necessary.
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 59
Number analyzed (Nasolabial Fold) | 118
score on a scale | -1.8 (0.6)

2. Primary Outcome: Proportion of Subjects With ≥1 Point Reduction in Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade Based on Investigator Assessment at Week 24
Description: The proportion of subjects with at least 1 point reduction from baseline in Nasolabial Folds-Severity Rating Scale (NLF-SRS) grade based on investigator assessment at week 24 after the initial treatment. The left and right nasolabial folds were graded separately. A subject is counted if the subject had at least one grade reduction over baseline on both nasolabial folds, on the 5-point NLF-SRS. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
Time Frame: Week 24
Population: The population consists of all participants who received the investigational device and had at least one post-treatment assessment (e.g., first pain assessment after injection).
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Participants | 58

3. Secondary Outcome: Change From Baseline in Average Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade Based on Investigator Assessment at Weeks 4 and 36
Description: Change from baseline in average Nasolabial Folds-Severity Rating Scale (NLF-SRS) grade based on investigator assessment at weeks 4 and 36 after the initial treatment. The left and right nasolabial folds were graded separately on the 5-point NLF-SRS then the average of the two sides was used for analysis. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
Time Frame: Baseline, Week 4, Week 36
Population: The population used consists of all participants who received the investigational device and had at least one post-treatment assessment (e.g., first pain assessment after injection). Only subjects with available data for the respective visit were included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Nasolabial Fold
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 59
Number analyzed (Nasolabial Fold) | 118
score on a scale
  Week 4 | -1.98 (0.4)
  Week 36 | -1.67 (0.61)

4. Secondary Outcome: Proportion of Subjects With ≥1 Point Reduction in Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade Based on Investigator Assessment at Weeks 4 and 36
Description: The proportion of subjects with at least 1 point reduction from baseline in Nasolabial Folds-Severity Rating Scale (NLF-SRS) grade based on investigator assessment at weeks 4 and 36 after the initial treatment. The left and right nasolabial folds were graded separately. A subject is counted if the subject had at least one grade reduction over baseline on both nasolabial folds, on the 5-point NLF-SRS. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
Time Frame: Week 4, Week 36
Population: The population used consists of all participants who received the investigational device and had at least one post-treatment assessment (e.g., first pain assessment after injection).
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Participants
  Week 4 | 59
  Week 36 | 58

5. Secondary Outcome: Proportion of Subjects With Aesthetic Improvement Based on Investigator Assessment at Weeks 4, 24 and 36
Description: The proportion of subjects with an aesthetic improvement over baseline (subjects who have been rated as "very much improved" or "much improved" or "improved" on both nasolabial folds), based on investigator assessment at weeks 4, 24 and 36 after the initial treatment and using the 5-point Global Aesthetic Improvement Scale (GAIS). GAIS grades are ranked as "very much improved", "much improved", "improved", "no change", and "worse".
Time Frame: Week 4, Week 24, Week 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Participants
  Week 4 | 59
  Week 24 | 59
  Week 36 | 58

6. Secondary Outcome: Satisfaction of Subjects With Aesthetic Outcome at Weeks 4, 24 and 36
Description: Summary of subjects' satisfaction with aesthetic outcome of the treatment at weeks 4, 24 and 36 after the initial treatment. Subjects were asked to rate their satisfaction with the treatment using one of the following categories: 'very unsatisfied', 'unsatisfied', 'neither unsatisfied nor satisfied', 'satisfied', or 'very satisfied'.
Time Frame: Week 4, Week 24, Week 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Participants
  Week 4: Unsatisfied | 1
  Week 4: Neither unsatisfied nor satisfied | 2
  Week 4: Satisfied | 5
  Week 4: Very satisfied | 51
  Week 4: Missing | 1
  Week 24: Unsatisfied | 2
  Week 24: Neither unsatisfied nor satisfied | 1
  Week 24: Satisfied | 9
  Week 24: Very satisfied | 47
  Week 24: Missing | 1
  Week 36: Unsatisfied | 0
  Week 36: Neither unsatisfied nor satisfied | 3
  Week 36: Satisfied | 7
  Week 36: Very satisfied | 49
  Week 36: Missing | 1

7. Secondary Outcome: Average Pain Intensity Based on Subject Assessment Immediately After the Last Injection and 15 Minutes Thereafter for Initial and Touch-up Treatment
Description: Average pain intensity based on subject assessment immediately after the last injection and about 15 minutes thereafter for initial treatment at baseline and for touch-up treatment at week 2 (if applicable). Subjects quantified the pain associated with the procedure using a semi-quantitative 11-point Numeric Pain Rating Scale (NPRS): 0 is no pain and 10 is the worst pain you can imagine.
Time Frame: Baseline - Immediately after end of treatment, 15 minutes after end of treatment Week 2 - Immediately after end of treatment, 15 minutes after end of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
score on a scale
  Pain assessment immediately after end of treatment - Baseline | 1.5 (1.4)
  Pain assessment 15 minutes after end of treatment - Baseline | 0.0 (0.0)
  Pain assessment immediately after end of treatment - Week 2: number analyzed (Participants) | 20
  Pain assessment immediately after end of treatment - Week 2 | 2.1 (1.8)
  Pain assessment 15 minutes after end of treatment - Week 2: number analyzed (Participants) | 20
  Pain assessment 15 minutes after end of treatment - Week 2 | 0.0 (0.0)

8. Secondary Outcome: Proportion of Subjects With ≥1 Point Reduction in Nasolabial Folds-Severity Rating Scale (NLF-SRS) Grade Based on Independent Reviewer Assessment of Photographs at Week 24
Description: The proportion of subjects with at least 1 point reduction from baseline in Nasolabial Folds-Severity Rating Scale (NLF-SRS) grade based on independent reviewer assessment of photographs at week 24 after the initial treatment. The left and right nasolabial folds were graded separately. A subject is counted if the subject had at least one grade reduction over baseline on both nasolabial folds, on the 5-point NLF-SRS. NLF-SRS scores are ranked as 0 (None/minimal), 1 (Mild), 2 (Moderate), 3 (Severe) and 4 (Extreme).
Time Frame: Week 24
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® FILLER Lidocaine
Number analyzed (Participants) | 60
Participants | 59

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Princess® FILLER Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60
Other Adverse Events (participants affected / at risk) | 27/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Princess® FILLER Lidocaine (N=60)
Haematoma infection (Infections and infestations) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Princess® FILLER Lidocaine (N=60)
Lip haematoma (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Injection site haematoma (General disorders) | 16 (17)
Injection site pain (General disorders) | 12 (12)
Injection site swelling (General disorders) | 2 (2)
Periodontitis (Infections and infestations) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03611491/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03611491/SAP_001.pdf